CLINICAL TRIAL: NCT00659009
Title: The Effects of Mild Hypobaric Hypoxia on Oxygen Saturation During Sleep: An Investigation of the Physiologic Mechanisms and Significance
Brief Title: Effects of Mild Hypobaric Hypoxia on Oxygen Saturation During Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Boeing Company (Industry)
Collaborators: Simon Fraser University (Other); Massey University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Boeing-003
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2010-02

CONDITIONS: Sleep-related Respiratory Disturbance
Keywords: environmental; hypobaric hypoxia; sleep; respiratory-disturbance; neurobehavioral performance; Effect of altitude on sleep-related respiratory disturbance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Barometric pressure equivalent to sea level (760 mm Hg).
  Interventions: Other: Sea level equivalent barometric pressure
- 2 (Experimental): Barometric pressure equivalent to 6000 feet (609 mm Hg)
  Interventions: Other: Reduced barometric pressure
- 3 (Experimental): Barometric pressure equivalent to 8000 feet (565 mm Hg).
  Interventions: Other: Reduced barometric pressure

INTERVENTIONS:
Other: Reduced barometric pressure — Sleep in reduced barometric pressure environment.
  Arms: 2
Other: Sea level equivalent barometric pressure — Sleep in barometric pressure equivalent to sea level.
  Arms: 1
Other: Reduced barometric pressure — Sleep in reduced barometric pressure environment.
  Arms: 3

SUMMARY:
Ascent to altitude lowers oxygen saturation. In addition, sleep lowers oxygen saturation at any altitude. In a prior study, we observed that sleep at 8000 feet resulted in pronounced reduction in oxygen saturation, but did not result in reduced post sleep neurobehavioral performance or impaired sleep quality or quantity. We plan to do a more sophisticated physiological evaluation of the respiratory mechanisms responsible for the reduced oxygen saturation and determine if there are any adverse consequences to this level of intermittent hypoxia. We anticipate that central respiratory apnea is the physiologic mechanism, and that there will not be persistent changes in autonomic nervous activity measured by heart rate variability.

DETAILED DESCRIPTION:
This study has 6 primary objectives/hypotheses:

1. Replicate findings of earlier study in which no effects of altitude were observed on post sleep neurobehavioral performance, sleep quantity or quality.
2. Determine if sleep at 6000 feet has effects similar to sleep at 8000 feet.
3. Identify if central or obstructive apnea is responsible for the reduction in oxygen saturation observed during sleep at 8000 feet.
4. Determine if respiratory abnormalities observed at 6000 feet are similar but less severe than at 8000 feet.
5. Determine if there are individual differences in respiratory physiology at sea level that enable prediction of pronounced respiratory disturbances during sleep at altitude.
6. Determine if changes in autonomic nervous activity, measured by heart rate variability, occur, and if so, do they persist for 8 hours.

Twenty healthy males between 30 and 60 years of age whose baseline apnea-hypopnea index is less than 15/hour will be recruited from the general population surrounding Burnaby, British Columbia, Canada. Women are excluded because of the changes in sleep structure associated with the menstrual cycle.

Participants will be involved in the blinded crossover study for a 14 day period during which time they will monitor their sleep by actigraphy and sleep diaries, will spend 2 nights an altitude chamber at Simon Fraser University at ambient barometric pressure to become adapted to sleeping in that environment, then spend 3 study nights, each followed by 2 rest nights, sleeping at barometric pressures equivalent to sea level, 6000 feet, and 8000 feet. The order of exposures will be randomly balanced.

Pre study physiologic measures will include hypoxic ventilatory response, hypercapnic ventilatory response, and during one of the adaptation nights, apnea hypoxia index. Study sessions will consist of a 4 hour presleep period, a 6 hour sleep period, and a 1 hour post sleep period at the study barometric pressure. During the study sessions, heart rate, SpO2, polysomnographic measures, nasal air flow rates, and chest motion will be monitored and recorded. Psychomotor Vigilance Task response time will be measured before and after the sleep period. Heart rate will be recorded by ambulatory recording equipment for 8 hours following return to ambient barometric pressure conditions. This will be analyzed to determine if changes in heart rate variability are persistent.

Outcomes of primary interest will include total sleep time, duration of sleep stages, oxygen saturation, heart rate and heart rate variability, respiratory rates, air flow, and chest motion to assess if central or obstructive apnea is temporally related to reductions in oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between 30 and 60 years of age.
* Healthy, able to pass FAA Class III examination
* Body mass index less than 30
* Height less than 75 inches
* Ability to read and speak English

Exclusion Criteria:

* Prolonged residence above 5000 feet
* Recent travel to altitudes above 5000 feet
* Use of drugs or medications that affect sleep
* History of mood or psychiatric disorders that affect sleep.
* History of medical conditions that increase risk of adverse effects of hypoxia.
* Apnea hypopnea index greater than 15/hr at ground level.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
SpO2 | Continuous during sleep
Respiratory Disturbance | Continuous during sleep
Sleep architecture | Continuous during sleep

SECONDARY OUTCOMES:
Heart rate variability | Continuous during sleep and 8 hr following exposure

CONTACTS AND LOCATIONS:
Overall Officials: James M Muhm, MD, MPH, Principal Investigator — The Boeing Company
Locations (1):
- Environmental Physiology Unit, School of Kinesiology, Simon Fraser University, Burnaby, British Columbia, Canada